CLINICAL TRIAL: NCT00002476
Title: Phase III Randomized Study of Radiotherapy Alone vs With Concurrent Chemotherapy With MTX or VBMF (VCR/BLEO/MTX/5-FU) vs Subsequent Chemotherapy vs Concurrent and Subsequent Chemotherapy in Patients With Advanced Head and Neck Cancer
Brief Title: Radiation Therapy With or Without Chemotherapy in Treating Patients With Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CRC-PHASE-III-91001; CDR0000076951 (Registry Identifier: PDQ (Physician Data Query)); UKHAN-1
Record Dates: First submitted 1999-11-01; First posted 2004-06-09 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2010-03

CONDITIONS: Head and Neck Cancer
Keywords: stage II squamous cell carcinoma of the lip and oral cavity; stage II verrucous carcinoma of the oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV verrucous carcinoma of the oral cavity; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Bleomycin; Fluorouracil; Leucovorin; Methotrexate; Vincristine; Radiotherapy

INTERVENTIONS:
Biological: bleomycin sulfate
Drug: fluorouracil
Drug: leucovorin calcium
Drug: methotrexate
Drug: vincristine sulfate
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET photon therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if radiation therapy plus chemotherapy is more effective than radiation therapy alone in treating patients with advanced head and neck cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy with or without chemotherapy in treating patients with advanced head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether the addition of methotrexate (MTX) or VBMF (vincristine/bleomycin/methotrexate/fluorouracil) to radiotherapy for advanced carcinoma of the head and neck (with or without primary surgery) influences locoregional control and prolongs survival. II. Determine whether an effect on locoregional control or survival is apparent when chemotherapy is given during or following radiotherapy and whether it is increased when chemotherapy is given at both times. III. Determine, in a special randomization of patients with cancer of the oral cavity or oropharynx, whether neck irradiation improves locoregional control and survival.

OUTLINE: Randomized study. Patients without prior surgery are randomized 1:2 to Arms I:II-IV, while those with prior surgery are randomized 1:1 between Arms I and II only. Patients with tumors of the oral cavity or oropharynx may elect additional randomization between Arms V and VI and will receive irradiation of the primary according to the Manchester regimen. Arm I: Radiotherapy. Irradiation of the primary and/or lymph nodes according to 1 of 2 regimens (Manchester 3-week schedule or SECOG 6-week schedule) using megavoltage equipment. Arm II: Radiotherapy plus Concurrent Single-agent or 4-Drug Combination Chemotherapy with Leucovorin Rescue. Involved-field irradiation as in Arm I; plus Methotrexate, MTX, NSC-740; with Leucovorin calcium, CF, NSC-3590; or VBMF: Vincristine, VCR, NSC-67574; Bleomycin, BLEO, NSC-125066; MTX; Fluorouracil, 5-FU, NSC-19893; with CF. Arm III: Radiotherapy plus Subsequent Single-agent or 4-Drug Combination Chemotherapy with Leucovorin Rescue. Involved-field irradiation as in Arm I; plus MTX or VBMF; with CF. Arm IV: Radiotherapy plus Concurrent and Subsequent Single-agent or 4-Drug Combination Chemotherapy with Leucovorin Rescue. Involved-field irradiation as in Arm I; plus MTX or VBMF; with CF. Arm V: Radiotherapy. Neck node irradiation using megavoltage equipment. Arm VI: Observation. No nodal irradiation.

PROJECTED ACCRUAL: At least 1,000 patients will be entered.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed squamous cell cancer of the head and neck suitable for treatment with radiotherapy T2, T3, or T4 primary lesions Any N No distant metastasis May also be anaplastic carcinoma, verrucous carcinoma, or transitional cell carcinoma (as of 1/97) No occult primaries (as of 1/97) No adenocarcinomas, lymphomas, or melanomas (as of 1/97) Synchronous head and neck tumors are eligible (tumor with the worse prognosis is entered into study) (as of 1/97) Patients receiving surgery to neck nodes only must be randomized as surgery patients (as of 1/97) Patients with tumors of the oral cavity or oropharynx may additionally elect randomization to nodal irradiation vs. no further therapy provided there is no second primary

PATIENT CHARACTERISTICS: Age: 75 and under for patients electing participation in the nodal vs. no nodal irradiation portion of the study Performance status: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Fit for any protocol treatment option Willing to receive any protocol treatment option Prior malignancy allowed provided the treating clinician considers the patient cured

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior therapy Chemotherapy: No prior therapy Endocrine therapy: No prior therapy Radiotherapy: No prior therapy Surgery: Prior biopsy or excision allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1990-01; Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Tobias, MD, Study Chair — University College London Hospitals
Locations (7):
- Raj Tilak, Indore, India
- United Kingdom (6):
  - Royal Sussex County Hospital, Brighton, England
  - Middlesex Hospital- Meyerstein Institute, London, England
  - Derriford Hospital, Plymouth, England
  - Southend General Hospital, Westcliff-on-Sea, England
  - Royal Victoria Hospital, Belfast, Northern Ireland
  - Belfast City Hospital Trust, Belfast, Northern Ireland

REFERENCES:
- [Result] Tobias JS, Monson K, Gupta N, Macdougall H, Glaholm J, Hutchison I, Kadalayil L, Hackshaw A; UK Head and Neck Cancer Trialists' Group. Chemoradiotherapy for locally advanced head and neck cancer: 10-year follow-up of the UK Head and Neck (UKHAN1) trial. Lancet Oncol. 2010 Jan;11(1):66-74. doi: 10.1016/S1470-2045(09)70306-7. Epub 2009 Oct 29. PMID 19875337